CLINICAL TRIAL: NCT03663920
Title: A Prospective Observational Cohort Study on HIV Infection and Risk Related Coinfections/Comorbidities in Indonesia
Brief Title: HIV Infection and Risk Related Coinfections/Comorbidities in Indonesia
Acronym: INAPROACTIVE
Status: Completed | Type: Observational
Sponsor: Ina-Respond (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: INA104; U1111-1263-2484 (Other: WHO UTN Number)
Record Dates: First submitted 2018-01-04; First posted 2018-09-10 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: HIV
Keywords: Viral Load; CD4; Mortality; Disease Progression
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects or subject's parent must be willing to allow storage plasma and buffy coat at baseline visit and plasma at every follow up visit. All samples will be stored at the INA-RESPOND Reference laboratory and at each site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
INA-PROACTIVE is a multicenter, prospective, observational cohort study of HIV positive antiretroviral-naïve and treatment-experienced individuals. No investigational treatment or intervention will be used by this study. All participants will be managed according to the Indonesian HIV/AIDS Treatment Guideline and/or the Standard of Care (SoC) in local clinical setting, with the addition of rapid HIV viral load, CD4 cell count and syphilis testing.

DETAILED DESCRIPTION:
This study will accept participants meeting the eligibility criteria and data will be collected at baseline visit and 6-monthly regular follow up visits for 3 years (at month 6, 12, 18, 24, 30, and 36). The study will allow a ± 3-month window period for each scheduled regular follow up visit to minimize loss to follow up. Additional follow up data may be collected between regular follow up visits on certain participants who meet the additional follow up criteria.

During each visit, data collection will include socio-demographics, family history, past and current medical history, clinical assessments, laboratory and/or other supporting diagnosis examination. Blood specimens from each study visits will be collected for future research on immune function, pathogenesis, and genetics or genomics of HIV and risk related coinfections/comorbidities. The stored specimens will be investigated during the study and/or after the study completion.

Based on the highest number of HIV cases in hospitals from the National HIV/AIDS Control Program (MoHRI, 2016), 33 hospitals were identified as the proposed study sites (Appendix B). Ten hospitals are established INA-RESPOND's study sites. They are Dr. Cipto Mangunkusumo Hospital, Prof. Dr. Sulianti Saroso Infectious Diseases Hospital, and Persahabatan Hospital in Jakarta; Dr. Hasan Sadikin Hospital, Bandung; Dr. Kariadi Hospital, Semarang; Dr. Sardjito Hospital, Yogyakarta; Dr. Soetomo Hospital, Surabaya; Sanglah Hospital, Denpasar; Dr. Wahidin Sudirohusodo Hospital, Makassar; and Kab. Tangerang Hospital, Banten.

Ten additional new study sites will be selected from the list (Appendix B) and the INA-RESPOND team will conduct site assessments to determine their willingness and readiness to be INA-PROACTIVE study sites. If site activation is lagging, other hospitals not on the list can also be assessed as a potential study sites.

The total 20 study sites will be activated gradually based on their readiness within 2 years (12 sites on year-1 and additional 8 sites on year-2). It is expected that the additional new sites will expand the network, increase participants' recruitment, and will be able to represent Indonesian situation.

ELIGIBILITY:
Inclusion criteria:

1. HIV positive by the Standard of Care.
2. Documented informed consent for participants' ≥18 years old or informed consent by parents/legally accepted representative (LAR) or assent for minor participants prior to study procedures.
3. Willing to comply with the study procedures.
4. Agrees to the collection and storage of specimens for use in future research on immune function, pathogenesis, and/or genetics/genomics of HIV and opportunistic infections. (The participant may decline participation in genetic or genomics research and will still be eligible for the study).

Exclusion criteria:

1. Plans to move away to an area where the participant will not be able to complete the study visits in 3 years.
2. Is currently imprisoned.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective descriptive study that aims to estimate the characteristics, including among death cases, of people living with HIV in Indonesia. The study population will include people living with HIV at any age, any sex/gender, any HIV-affected key populations, whether ART-naïve or treatment-experienced in Indonesia. To get an estimation with 95% confidence interval (95% CI) that represents the true value in population. We calculated the minimum death cases need to be observed using the proportion of female HIV patients among death cases in Indonesia in 2016 (31%) and case fatality rate for HIV patients in Indonesia, 2016 (1.11%). The minimum number of death to be observed and HIV patients to be enrolled
Sampling Method: Probability Sample
Enrollment: 4336 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of participants achieving viral suppression (HIV RNA Viral Load <1000 copies/mL) in Indonesia. | From date of enrollment until the date of 36 months of follow-up study visit, lost to follow-up or death, whichever came first, assessed up to 3 years
  Incidence of participants achieving viral suppression with HIV RNA Viral Load <1000 copies/mL.

SECONDARY OUTCOMES:
Proportion of participants with HIV RNA Viral Load <1000 copies/mL at baseline and every six-monthly follow-up visit. | From date of enrollment until the date of 36 months of follow-up study visit, lost to follow-up or death, whichever came first, assessed up to 3 years
  Proportion of participants with HIV RNA Viral Load <1000 copies/mL at baseline and every six-monthly follow-up visit as virological outcomes
Mean change in CD4+ cell count from baseline and every six-monthly follow-up visit. | From date of enrollment until the date of 36 months of follow-up study visit, lost to follow-up or death, whichever came first, assessed up to 3 years
  Evaluate the immunologic response by the CD4 measurement from baseline (Mean change in CD4+ cell count) and every six-monthly follow-up visit as immunological outcomes
Proportion of AIDS defining illnesses at baseline and every six-monthly follow-up visit. | From date of enrollment until the date of 36 months of follow-up study visit, lost to follow-up or death, whichever came first, assessed up to 3 years
  Proportion of AIDS defining illnesses from baseline and every six-monthly follow-up visit as disease progression outcomes
Proportion of serious non-AIDS disease at baseline and every six-monthly follow-up visit. | From date of enrollment until the date of 36 months of follow-up study visit, lost to follow-up or death, whichever came first, assessed up to 3 years
  Proportion of serious non-AIDS disease from baseline and every six-monthly follow-up visit as disease progression outcomes
Incidence of AIDS-related deaths at baseline and every six-monthly follow-up visit. | From date of enrollment until the date of 36 months of follow-up study visit, lost to follow-up or death, whichever came first, assessed up to 3 years
  Incidence of AIDS-related deaths at baseline and every six-monthly follow-up visit as the mortality outcomes
Incidence of non-AIDS-related deaths at baseline and every six-monthly follow-up visit. | From date of enrollment until the date of 36 months of follow-up study visit, lost to follow-up or death, whichever came first, assessed up to 3 years
  Incidence of non-AIDS-related deaths at baseline and every six-monthly follow-up visit as the mortality outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. dr. Tuti Parwati Merati, Sp.PD.KPTI, Principal Investigator — Faculty of Medicine Udayana University-Sanglah Hospital, Denpasar
Locations (19):
- Indonesia (19):
  - Site 520: University of Udayana/Sanglah Hospital, Denpasar, Bali
  - Site 560: University of Diponegoro/ Dr. Kariadi Hospital, Semarang, Central of Java
  - Site 530: University of Indonesia/ Dr. Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta
  - Site 540: Penyakit Infeksi Sulianti Saroso Hospital, Jakarta, DKI Jakarta
  - Site 590: Persahabatan Hospital, Jakarta, DKI Jakarta
  - Site 660 RSUD Abdul Wahab Sjahranie, Samarinda, East Kalimantan
  - Site 700 - RSUD Dr.TC Hillers, Maumere, East Nusa Tenggara
  - Site 570: University of Airlangga/ Dr. Soetomo Hospital, Surabaya, East of Java
  - Site 600 : Adam Malik Hospital, Medan, North Sumatra
  - Site 650: Budi Kemuliaan Hospital, Batam, Riau Islands
  - Site 630: M. Ansari Saleh Hospital, Banjarmasin, South Kalimantan
  - Site 690 - RSUD Abepura, Jayapura, Special Region of Papua
  - Site 510: University of Padjajaran/ Dr. Hasan Sadikin Hospital, Bandung, West Java
  - Site 610 : RSU Kabupaten Tangerang, Tangerang, West Java
  - Site 680 - RSUD dr Soedarso, Pontianak, West Kalimantan
  - Site 670 - RSUD Dr. Zainoel Abidin, Banda Aceh
  - Site 640: St. Carolus Hospital, Jakarta
  - Site 550: University of Hassanudin/ Dr. Wahidin Sudirohusodo Hospital, Makassar
  - Site 580: University of Gadjah Mada/ Dr. Sardjito Hospital, Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merati TP, Yunihastuti E, Wisaksana R, Kurniati N, Arlinda D, Karyana M, Susanto NH, Lokida D, Kosasih H, Diana A, Bang LE, Setiyaningrum M, Amin DM, Eppy E, Cahyawati WASN, Danudirgo EW, Darmaja IMG, Farhanah N, Gunawan CA, Hadi U, Jamil KF, Katu S, Kembaren T, Kosa IGR, Norosingomurti DL, Purnama A, Laksanawati IS, Rusli A, Somia IKA, Subronto YW, Toruan IL, Ridzon R, Liang CJ, Neal AT, Chen RY; INA-PROACTIVE Study Group. A prospective observational cohort study of HIV infection in Indonesia: baseline characteristics and one-year mortality. BMC Infect Dis. 2025 Jan 20;25(1):87. doi: 10.1186/s12879-024-10354-8. PMID 39833697